CLINICAL TRIAL: NCT03756233
Title: Gradual Withdrawal of Remifentanil Infusion Reduced Postoperative Pain and Opioid Requirement During Breast Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: SMC2018-07-153
Record Dates: First submitted 2018-10-25; First posted 2018-11-28 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2018-10

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Remifentanil

STUDY DESIGN:
Intervention Model Description: In this study, remifentanil gradually withdrawal goup (test group) and remifentanil immediately stop group (control group) were divided into two groups. In the Remifentanil gradual reduction group (test group), 20 minutes before the end of the operation, remifentanil was gradually decreased by 25% every 5 minutes. The control group stopped remifentanil 10 minutes before the end of the operation.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remifentanil gradually withdrawal group (Active Comparator): 20 minutes before the end of the operation, remifentanil was gradually decreased by 25% every 5 minutes.
  Interventions: Drug: Remifentanil
- Remifentanil immediately stop group (Active Comparator): The control group stopped remifentanil 10 minutes before the end of the operation.
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — Remifentanil is a potent, short-acting synthetic opioid analgesic drug. It is given to patients during surgery to relieve pain and as an adjunct to an anesthetic.

SUMMARY:
Although remifentanil provides profound analgesia during operation, postoperative occurrence of hyperalgesia and tolerance after remifentanil administration could be a challenge to the postoperative pain control. Evaluation of analgesia and anti-nociception during anesthesia is still a challenging issue. Surgical Pleth Index (SPI) is a non-invasive and simple access tool used to monitor autonomous nervous system during anesthesia. This technique is based on photoplethysmographic wave and heart beat analysis. SPI values range between 0 (no stress) and 100 (high stress level). The purpose of this study was to determine the appropriate use of Remifentanil for pain control in patients with SPI.

DETAILED DESCRIPTION:
Patients were randomized into either SPI-guided analgesia or standard practice (Control). In both groups, anesthesia was maintained with total intravenous anaesthesia(TIVA) to keep bispectral index values between 40 and 60.

In the Remifentanil gradual reduction group (test group), 20 minutes before the end of the operation, remifentanil was gradually decreased by 25% every 5 minutes. The control group stopped remifentanil 10 minutes before the end of the operation.

SPI was recorded before the intubation, after the intubation, directly before the end of surgery. The number of unwanted somatic events, hemodynamics, Patient-controlled analgesia(PCA) consumption, narcotic analgesics consumption, and recovery times were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received the breast conserving surgery

Exclusion Criteria:

* Patients with arrhythmia who have poor SPI measurement
* When the patient refused
* Patients with decreased renal function of Cr> 2
* Surgery for more than 3 hours, surgery expected to bleed more than 500 ml

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-03 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale(NRS) | postoperative 1 hour
  The difference of postoperative highest pain score (NRS) between two groups

SECONDARY OUTCOMES:
SPI | intraoperative (after the laryngeal mask airway)
  The difference of Surgical Pleth Index between two groups
SPI | intraoperative (after the incision)
  The difference of Surgical Pleth Index between two groups
analgesics consumption | during post-anesthesia care unit
  The difference of analgesics consumption between two groups
analgesics consumption | up to postoperative 48hours
  The difference of analgesics consumption between two groups
nausea & vomiting | postoperative 1 hour
  The difference of nausea and vomiting between two groups
Numeric Rating Scale(NRS) | during postoperative 48hours
  The difference of highest postoperative pain score (NRS) between two groups
the duration of eye opening | end of surgery
  the duration of eye opening after stoping propofol
intraoperative remifentanil consumption | intraoperative
  the dose of intraoperative remifentanil according to postoperative pain

CONTACTS AND LOCATIONS:
Overall Officials: sehee kang, fellow, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Gangnam-gu, South Korea